CLINICAL TRIAL: NCT04831476
Title: A Non Interventional Post Authorisation Multicenter Study to Evaluate the Disease Control (Benign Prostate Hyperplasia Control) and Quality of Life (QoL) Following the 6-months Combination Treatment With Dutasteride and Tamsulosin. PROSPERITY Group of Studies (I&II).
Brief Title: Α Prospective Observational Study for the Evaluation of Disease Control and Quality of Life in Patients With Benign PROStatic hyPERplasia Under Fixed Dose combΙnaTion Treatment With Dutasteride and Tamsulosin . PROSPERITY Group of Studies (I&II)
Acronym: PROSPERITY
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-DTM-EL-126/133
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-02

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostate Hyperplasia; IPSS (International Prostate Symptom Score); LUTS (Lower Urinary Tract Symptoms)
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with Benign Prostate Hyperplasia — patients with benign prostatic hyperplasia under fixed dose combΙnation treatment with dutasteride and tamsulosin

SUMMARY:
Investigation of the efficacy and safety of the stable combination of dutasteride and tamsulosin (Dinaplex®) in the Greek population as well as the evaluation of the quality of life of patients with benign prostatic hyperplasia (BPH) in treatment with a stable combination of dutasteride and tamsulosin (Dinaplex®)

DETAILED DESCRIPTION:
Combination therapy with the 5-α reductase inhibitor, dutasteride, and the α-blocker, tamsulosin, in men with moderate to severe benign prostatic hyperplasia and prostate enlargement, was studied in the Combination of Avodart ™ and Tamsulosin (CombAT) which was a four-year, global, multicenter, randomized, double-blind, parallel design (3 arms) study. The aim of the study was to investigate the benefits of combination therapy (dutasteride-tamsulosin) compared to monotherapy in terms of improvement of symptoms and long-term results (AUR and surgery), in men with moderate to severe BPH. The primary endpoint in the two years since the start of the study was the change in the IPSS score, while the primary endpoint, after four years of treatment, was the time until the long-term results manifested (i.e. AUR or CF surgery) as well as the percentage of participants who were led to them. Patients were at least 50 years old with a prostate tumor ≥30 cm3 and a PSA level ≥ 1.5 ng / mL. 4838 men (39) participated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patient with moderate to severe BPH symptoms receiving either monotherapy, dual medication as monoproducts or other stable combination and not responding adequately to treatment.
* Adult male patient with BPH who has fully understood the study procedures and has signed a consent form after information.

Exclusion Criteria:

* Patient who does not meet the criteria for taking the study drug (s), according to the Summary of Product Characteristics of each drug in the study.

Ages: 18 Years to 85 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Adult males who based on physician's recommedations will receive
  DINAPLEX®- Each hard capsule contains 0.5 mg dutasteride and 0.4 mg tamsulosin hydrochloride (equivalent to 0.367 mg tamsulosin) Tamsulosin hydrochloride Tamsulosin binds selectively and competitively to postsynaptic α1A adrenergic receptors and to a lesser extent to α1D adrenergic receptors. It relaxes the smooth muscles of the prostate and urethra. By relaxing the smooth muscle fibers of the bladder sphincter, it relieves obstructive effects and increases urine flow. It has little antihypertensive effect.
  Doutasteride Dutasteride lowers circulating dihydrotestosterone (DHT) levels by inhibiting the 5a-reductase isoenzymes type I and II, which are responsible for converting testosterone to DHT. The effect of dutasteride on DHT levels is dose-dependent and is observed within 1-2 weeks (85% and 90% reduction respectively).
Sampling Method: Non-Probability Sample
Enrollment: 1296 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of disease control (BPH), PROSPERITY I Evaluation of quality of life. PROSPERITY II | 3-6 months
  The change in the overall score (questions 1-7) of the IPSS (International Prostate Symptom Score) questionnaire. PROSPERITY I.
  The change in the score of the question related to quality of life, of the IPSS questionnaire. PROSPERITY II

SECONDARY OUTCOMES:
Evaluation of disease control (BPH), PROSPERITY II. | 3-6 months
  The change in the overall score (questions 1-7) of the IPSS (International Prostate Symptom Score) questionnaire. PROSPERITY II.
U/S measurement. PROSPERITY I&II | 3-6 months
  The change in the volume of the prostate and the change in the volume of the remaining urine (measurement by ultrasound).
Number of AEs (PROSPERITY I&II) | 3-6 months
  The recording of Adverse Events (Adverse Events, SA) if they occur during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Laikon Hospital of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Medical Association Declaration of Helsinki. Ethical principles for Medical Research Involving Human Subjects, Helsinki 1964, amended in Tokyo 1975, Venice 1983, Hong Kong 1989, South Africa 1996, Edinburgh 2000, and Seoul 2008.
- [Result] Helga Fritch, Wolfgang Kühnel. Εγχειρίδιο Περιγραφικής Ανατομικής. s.l. : Π.Χ. Πασχαλίδης, 2009.
- [Result] Presti JC Jr. (2000) Neoplasms of the prostate gland, in Smith's General Urology, 15th Edition, Tanagho EA and McAninch JW, Editors. Lange Medical Books: New York, USA. p. 399-421.
- [Result] Shibata K, Hirasawa A, Moriyama N, Kawabe K, Ogawa S, Tsujimoto G. Alpha 1a-adrenoceptor polymorphism: pharmacological characterization and association with benign prostatic hypertrophy. Br J Pharmacol. 1996 Jul;118(6):1403-8. doi: 10.1111/j.1476-5381.1996.tb15552.x. PMID 8832064
- [Result] Ekman P. The prostate as an endocrine organ: androgens and estrogens. Prostate Suppl. 2000;10:14-8. No abstract available. PMID 11056488
- [Result] Verhamme KM, Dieleman JP, Bleumink GS, van der Lei J, Sturkenboom MC, Artibani W, Begaud B, Berges R, Borkowski A, Chappel CR, Costello A, Dobronski P, Farmer RD, Jimenez Cruz F, Jonas U, MacRae K, Pientka L, Rutten FF, van Schayck CP, Speakman MJ, Sturkenboom MC, Tiellac P, Tubaro A, Vallencien G, Vela Navarrete R; Triumph Pan European Expert Panel. Incidence and prevalence of lower urinary tract symptoms suggestive of benign prostatic hyperplasia in primary care--the Triumph project. Eur Urol. 2002 Oct;42(4):323-8. doi: 10.1016/s0302-2838(02)00354-8. PMID 12361895
- [Result] Jacobsen SJ, Jacobson DJ, Girman CJ, Roberts RO, Rhodes T, Guess HA, Lieber MM. Treatment for benign prostatic hyperplasia among community dwelling men: the Olmsted County study of urinary symptoms and health status. J Urol. 1999 Oct;162(4):1301-6. PMID 10492184
- [Result] Marberger MJ, Andersen JT, Nickel JC, Malice MP, Gabriel M, Pappas F, Meehan A, Stoner E, Waldstreicher J. Prostate volume and serum prostate-specific antigen as predictors of acute urinary retention. Combined experience from three large multinational placebo-controlled trials. Eur Urol. 2000 Nov;38(5):563-8. doi: 10.1159/000020356. PMID 11096237
- [Result] Clifford GM, Logie J, Farmer RD. How do symptoms indicative of BPH progress in real life practice? The UK experience. Eur Urol. 2000;38 Suppl 1:48-53. doi: 10.1159/000052401. PMID 11111208
- [Result] Lowe FC. Goals for benign prostatic hyperplasia therapy. Urology. 2002 Feb;59(2 Suppl 1):1-2. doi: 10.1016/s0090-4295(01)01554-0. No abstract available. PMID 11832306
- [Result] Sanda MG, Beaty TH, Stutzman RE, Childs B, Walsh PC. Genetic susceptibility of benign prostatic hyperplasia. J Urol. 1994 Jul;152(1):115-9. doi: 10.1016/s0022-5347(17)32831-8. PMID 7515446
- [Result] Sidney S, Quesenberry CP Jr, Sadler MC, Guess HA, Lydick EG, Cattolica EV. Incidence of surgically treated benign prostatic hypertrophy and of prostate cancer among blacks and whites in a prepaid health care plan. Am J Epidemiol. 1991 Oct 15;134(8):825-9. doi: 10.1093/oxfordjournals.aje.a116157. PMID 1719806
- [Result] Choi J, Ikeguchi EF, Lee SW, Choi HY, Te AE, Kaplan SA. Is the higher prevalence of benign prostatic hyperplasia related to lower urinary tract symptoms in Korean men due to a high transition zone index? Eur Urol. 2002 Jul;42(1):7-11. doi: 10.1016/s0302-2838(02)00222-1. PMID 12121722
- [Result] Geller J, Sionit L, Partido C, Li L, Tan X, Youngkin T, Nachtsheim D, Hoffman RM. Genistein inhibits the growth of human-patient BPH and prostate cancer in histoculture. Prostate. 1998 Feb 1;34(2):75-9. doi: 10.1002/(sici)1097-0045(19980201)34:23.0.co;2-i. PMID 9465938
- [Result] Chyou PH, Nomura AM, Stemmermann GN, Hankin JH. A prospective study of alcohol, diet, and other lifestyle factors in relation to obstructive uropathy. Prostate. 1993;22(3):253-64. doi: 10.1002/pros.2990220308. PMID 7683816
- [Result] Ryl A, Rotter I, Miazgowski T, Slojewski M, Dolegowska B, Lubkowska A, Laszczynska M. Metabolic syndrome and benign prostatic hyperplasia: association or coincidence? Diabetol Metab Syndr. 2015 Oct 29;7:94. doi: 10.1186/s13098-015-0089-1. eCollection 2015. PMID 26516352
- [Result] Peters TJ, Donovan JL, Kay HE, Abrams P, de la Rosette JJ, Porru D, Thuroff JW. The International Continence Society "Benign Prostatic Hyperplasia" Study: the botherosomeness of urinary symptoms. J Urol. 1997 Mar;157(3):885-9. PMID 9072592
- [Result] Scarpa RM. Lower urinary tract symptoms: what are the implications for the patients? Eur Urol. 2001;40 Suppl 4:12-20. doi: 10.1159/000049890. PMID 11786675
- [Result] Garraway WM, Collins GN, Lee RJ. High prevalence of benign prostatic hypertrophy in the community. Lancet. 1991 Aug 24;338(8765):469-71. doi: 10.1016/0140-6736(91)90543-x. PMID 1714529
- [Result] Lepor H. Alpha 1-adrenoceptor selectivity: clinical or theoretical benefit? Br J Urol. 1995 Jul;76 Suppl 1:57-61. No abstract available. PMID 7544216
- [Result] Welch G, Kawachi I, Barry MJ, Giovannucci E, Colditz GA, Willett WC. Distinction between symptoms of voiding and filling in benign prostatic hyperplasia: findings from the Health Professionals Follow-up Study. Urology. 1998 Mar;51(3):422-7. doi: 10.1016/s0090-4295(97)00626-2. PMID 9510347
- [Result] International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use.. ICH harmonized tripartite guideline: Guideline for Good Clinical Practice. J Postgrad Med. 2001 Jan-Mar;47(1):45-50. No abstract available. PMID 11590294
- [Result] Epstein M; International Society of Pharmacoepidemiology. Guidelines for good pharmacoepidemiology practices (GPP). Pharmacoepidemiol Drug Saf. 2005 Aug;14(8):589-95. doi: 10.1002/pds.1082. No abstract available. PMID 15918159